CLINICAL TRIAL: NCT06549335
Title: The Efficacy and Safety of Zanubrutinib, Obinutuzumab and Lenalidomide (ZGR) Regimen in High-risk Treatment-naive Patients with Follicular Lymphoma
Brief Title: Zanubrutinib, Obinutuzumab and Lenalidomide (ZGR) in High-risk Treatment-naive Patients with Follicular Lymphoma (FL)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL-ZGR
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Follicular Lymphoma
Keywords: Zanubrutinib; Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — zanubrutinib; obinutuzumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Zanubrutinib, Obinutuzumab and Lenalidomide (ZGR) (Experimental)
  Interventions: Drug: Zanubrutinib, Obinutuzumab and Lenalidomide (ZGR)

INTERVENTIONS:
Drug: Zanubrutinib, Obinutuzumab and Lenalidomide (ZGR) — Induction therapy:
  The ZGR regimen will be given from day 1 of each cycle of treatment. Each cycle will last for 28 days. Participants will receive a total of 6 cycles.
  Dosage:
  1. Zanubrutinib, 160 mg bid, po, day 1-28;
  2. Obinutuzumab, 1000mg, ivgtt, day 1/8/15 (C1), day1 (C2-6);
  3. Lenalidomide, 25 mg qd, po, day 2-11.
  Maintenance therapy:
  1. Obinutuzumab, ivgtt,1000mg, every 3 months for 2 years;
  2. Lenalidomide, 25mg, PO, during 1-10 days in every 28 days for 6 cycles.

SUMMARY:
This is a prospective, multiple-centers, open-label, single-arm clinical study designed to evaluate the efficacy and safety of Zanubrutinib, Obinutuzumab, and Lenalidomide (ZGR) in high-risk treatment-naive patients with follicular lymphomas

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed CD20 positive follicular lymphoma grade 1, 2, or 3A based on 2016 WHO classification
2. Treatment naive
3. Age ≥ 18 years
4. Indications for treatment confirmed
5. Identified as high-risk group by Follicular Lymphoma International Prognostic Index 2 (FLIPI2) at enrollment
6. Must has measurable lesion in CT or PET-CT prior to treatment
7. Considered suitable for ZGR regimens
8. Informed consented

Exclusion Criteria:

* Transformed follicular lymphoma or 3B follicular lymphoma;
* HBsAg positive and / or HBcAb positive with HBV DNA titer; HCV antibody positive with HCV-RNA; or HIV positive
* Any drug contraindication in the treatment plan
* Pregnant or lactating women
* Patients judged by other researchers to be unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At the end of Cycle 6 (each cycle is 28 days)
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Complete response rate (CR) | At the end of Cycle 6 (each cycle is 28 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Partial response rate (PR) | At the end of Cycle 6 (each cycle is 28 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Duration of response | Baseline up to data cut-off (up to approximately 2 years)
  Time from first occurrence of documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR. Tumor assessments were performed with PET-CT.
2-year progression free survival rate | Baseline up to data cut-off (up to approximately 2 years)
  progression-free survival was defined as the time from the date of first treatment until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
2-year overall survival rate | Baseline up to data cut-off (up to approximately 2 years)
  progression-free survival was defined as the time from the date of first treatment until the date of the first documented day of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No